CLINICAL TRIAL: NCT06545110
Title: Retinol Binding Protein 4 Expression and Its Genetic Variants in Severe Alopecia Areata Treated With Barcitinib.
Brief Title: Retinol Binding Protein 4 Protein in Alopecia Areata Treated With Barcitinib
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Marwa Alyan Abd-elaziz Mohammed, assistant lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBP4 in alopecia areata
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Alopecia Areata
Keywords: Retinol binding protein 4 , Barcitinib
MeSH Terms: conditions — Alopecia Areata | interventions — baricitinib

STUDY DESIGN:
Who Masked: Investigator
Masking Description: asses level of retinol binding protein 4 before and after barcitinib treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): 60 patient with sever alopecia areata
  Interventions: Drug: Baricitinib Oral Tablet
- group B (Placebo Comparator): 60 healthy individuals
  Interventions: Drug: Baricitinib Oral Tablet

INTERVENTIONS:
Drug: Baricitinib Oral Tablet — Baricitinib 2/4mg giving to patients with sever alopecia areata after assessment Retinol Binding Protein 4 and its genetic variations.

SUMMARY:
Assess serum and tissue retinol binding protein 4 in patients with severe alopecia areata in correlation with healthy individuals .

Estimate genetic profile of retinol binding protein4 in severe alopecia areata patients

Assess possible role of retinol binding protein 4 genetic mutation in response to barcitinib treatment in patients with severe alopecia areata .

DETAILED DESCRIPTION:
Alopecia areata is an autoimmune disorder characterized by transient, non-scarring hair loss and preservation of the hair follicle .It is a multifactorial disease in which environmental, neuro-endocrinological, immunological and genetic factors are involved . AA affecting the hair follicle is the most common form, through a breakdown in immune privilege of the hair follicle in the anagen (hair growth) phase by CD4+ and CD8+ T lymphocytes .

Based on the degree of hair loss and variation in clinical presentation, AA classified into patchy (AA; localized areas of hair loss on the scalp and/or body), totalis (AT; entire scalp hair loss), and universalis (AU; entire scalp and body hair loss . Several studies showed that genes involved in immune response , inflammatory diseases . infectious diseases .The hair loss in AA involves changes in the hair growth cycle, resulting in dystrophic anagen hair follicles together with increased frequency of telogen follicles.

Retinol binding protein 4 (RBP4) is a member of the lipocalin family and the major transport protein of the hydrophobic molecule retinol, also known as vitamin A, in the circulation. Expression of RBP4 is highest in the liver, where most of the body's vitamin A reserves are stored as retinyl esters. For the mobilization of vitamin A from the liver, retinyl esters are hydrolyzed to retinol, which then binds to RBP4 in the hepatocyte . The pathogenesis of AA may be related to increased serum retinol-binding protein-4 (RBP4) level. Its level was found to be increasing in the outer root sheath during late anagen and remained as such throughout catagen. RBP4 may contribute to inflammation by stimulating the expression of proinflammatory molecules involved in leukocyte recruitment and adherence to the endothelium .

Baricitinib (bar" i sye' ti nib) is an orally available, specific inhibitor Janus-associated kinases (mainly JAK1 and JAK2) that is used to treat moderate-to-severe rheumatoid arthritis and alopecia areata. The Janus kinases are critical steps in immune activation as well as in hematopoiesis. JAK1 is a critical kinase in the cellular responses of interferon alpha while JAK2 is involved in pathways activated by interferon gamma. The immunomodulatory effects of baricitinib have led to its evaluation in several autoimmune conditions interrupt cytokine signaling implicated in the pathogenesis of alopecia areata .

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 12 years old not more than 60 with severe alopecia areata, multiple or /with not responding to usual treatment

Exclusion Criteria:

* Patients with scarring alopecia.
* Patients less than 12 years old or more than 60.
* Patients with active inflammatory disease or immuncompromised.
* Patients with infection or malignancy .
* Patients with antiepileptic drugs or psychotics .
* Pregnancy and lactation .
* Patients with abnormal lipid profile.
* Patients with bleeding or thrombotic tendency.
* Patients taking other JAK inhibitors or cyclosporine or immunosuppressive drugs.
* Patients with active herpes zoster or have tendency for recurrence.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Assess serum and tissue retinol binding protein 4 in patients with severe alopecia | baseline
  Assess serum and tissue retinol binding protein 4 in patients with severe alopecia in serum and tissue samples in response to Baricitinib .

SECONDARY OUTCOMES:
Estimate genetic profile of retinol binding protein4 in severe alopecia areata patients | baseline
  Estimate genetic variations of Retinol binding protein 4 in blood samples before and after Baricitinib.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Adam Ali El Tieb, professor, Study Director — Aswan University; Mohamed Hosny Hassan, professor, Study Director — South Valley University; Eisa Mohammed Hegazy, professor, Study Director — South Valley University
Locations (1):
- South Valley University, Qina, الكيلو 6 Qena - Safaga Rd, Qena, Qena Governorate, Egypt

REFERENCES:
- [Background] King B, Ohyama M, Kwon O, Zlotogorski A, Ko J, Mesinkovska NA, Hordinsky M, Dutronc Y, Wu WS, McCollam J, Chiasserini C, Yu G, Stanley S, Holzwarth K, DeLozier AM, Sinclair R; BRAVE-AA Investigators. Two Phase 3 Trials of Baricitinib for Alopecia Areata. N Engl J Med. 2022 May 5;386(18):1687-1699. doi: 10.1056/NEJMoa2110343. Epub 2022 Mar 26. PMID 35334197
- [Background] Steinhoff JS, Lass A, Schupp M. Biological Functions of RBP4 and Its Relevance for Human Diseases. Front Physiol. 2021 Mar 11;12:659977. doi: 10.3389/fphys.2021.659977. eCollection 2021. PMID 33790810
- [Background] Al-Eitan LN, Alghamdi MA, Al Momani RO, Aljamal HA, Abdalla AM, Mohammed HM. Genetic predisposition of alopecia areata in jordanians: A case-control study. Heliyon. 2022 Mar 24;8(4):e09184. doi: 10.1016/j.heliyon.2022.e09184. eCollection 2022 Apr. PMID 35392398
- [Background] Bhardwaj P, Basu D, Podder I, Gharami RC. Clinico-Epidemiological Profile of Childhood Alopecia Areata Along with Dermoscopic Correlation: A Cross-Section, Observational Study. Indian Dermatol Online J. 2021 Mar 2;12(2):250-257. doi: 10.4103/idoj.IDOJ_451_20. eCollection 2021 Mar-Apr. PMID 33959521
- [Background] Gil-Quinones SR, Sepulveda-Pachon IT, Sanchez Vanegas G, Gutierrez-Castaneda LD. Effect of PTPN22, FAS/FASL, IL2RA and CTLA4 genetic polymorphisms on the risk of developing alopecia areata: A systematic review of the literature and meta-analysis. PLoS One. 2021 Nov 4;16(11):e0258499. doi: 10.1371/journal.pone.0258499. eCollection 2021. PMID 34735462
- [Background] Pratt CH, King LE Jr, Messenger AG, Christiano AM, Sundberg JP. Alopecia areata. Nat Rev Dis Primers. 2017 Mar 16;3:17011. doi: 10.1038/nrdp.2017.11. PMID 28300084